CLINICAL TRIAL: NCT01853436
Title: Impact of Acellular Dermal Matrix in Reduction of Surgical Complexity of Breast Reconstructions With Implants
Brief Title: Impact of ADM in Reduction of Surgical Complexity of Breast Reconstructions With Implants (Nava)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lifecell became part of Allergan; company deciscion
Sponsor: LifeCell (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LFC 2012.04.01
Record Dates: First submitted 2013-05-07; First posted 2013-05-15 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Patients With Breast Cancer Requiring Mastectomy and Suitable for Reconstruction
Keywords: Breast Cancer; Reconstructive Tissue Matrix; Acellular Dermal Matrices (ADM)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single stage reconstructions (Experimental): as defined for use in the Experimental arm
  Interventions: Device: Strattice™ Reconstructive Tissue Matrix
- Two stage breast reconstructions (Other): CONTROL: standard two stage breast reconstructions without Acellular dermal matrices (ADM), in patients who are clinically suitable candidates for reconstruction with Acellular dermal matrices(ADM)based single stage reconstruction technique. Reconstructions with Strattice™ Reconstructive Tissue Matrix
  Interventions: Device: Strattice™ Reconstructive Tissue Matrix

INTERVENTIONS:
Device: Strattice™ Reconstructive Tissue Matrix — Experimental arm: Device: Strattice Reconstructive Tissue Matrix Unilateral or bilateral mastectomy. Immediate breast reconstruction with sub-pectoralis muscle placement of a breast implant with ADM, single stage reconstruction technique. Control arm: Device: no device. Immediate breast tissue expander/implant based reconstruction with a two-stage reconstruction technique.

SUMMARY:
The objective of this study is to demonstrate that acellular dermal matrix, Strattice™ Reconstructive Tissue Matrix, can reduce the surgical complexity and post-operative pain of breast reconstructions with implants by avoiding one more surgical step in the operating room.

DETAILED DESCRIPTION:
This study is designed to compare the clinical outcomes of patients undergoing mastectomy followed by a direct to implant breast reconstruction with Strattice™ Reconstructive Tissue Matrix to patients undergoing a standard two-stage reconstruction without Strattice™ or any other mesh or tissue flap.

Potential candidates for the study will be identified through routine practice. Women who meet the inclusion and exclusion criteria will be invited to participate in the study. A screening visit will take place maximally 30 days prior to surgery.

Randomization will occur maximally 7 days prior to the mastectomy procedure. As some women may have to undergo bilateral mastectomy and reconstruction, the randomization scheme will ensure that both breasts will be reconstructed with the same surgical approach.

The Day of Surgery consists of both a mastectomy and a breast reconstruction. The surgical site and the breasts will be evaluated on the day of hospital discharge and at postoperative days 14 and 30 for all patients after each hospital admission. During these visits, the breasts will be examined and an Acute Inflammatory Assessment (AIR) will be completed. In addition the breast flaps and incisions will be evaluated for signs of infection, seroma, hematoma or skin necrosis.

ELIGIBILITY:
Inclusion Criteria:

A study patient may be included if she:

1. Has planned to undergo a unilateral or bilateral mastectomy and have small to medium size breasts (predicted breast implant size maximally 500 gms), with none or moderate (Grade 1 or 2) ptosis, and healthy, sufficiently thick, well-vascularized skin flaps anticipated by the surgeon.
2. Is a clinically suitable candidate for immediate reconstruction with ADM based single stage reconstruction technique (as defined for use in the Experimental arm).
3. Is female, ≥18 years of age.
4. Is willing to undergo immediate breast reconstruction with sub-pectoralis muscle placement of a breast implant by either the Experimental (ADM based single stage) or the Control (TE/Implant based two stage) techniques.
5. Is in good health other than breast pathology and is suited to general anesthesia and planned treatments.
6. Understands and is willing to follow all aspects of the study protocol including randomization and has signed and dated the approved Informed Consent Form prior to any study-related procedures being performed.

Exclusion Criteria:

A study patient is excluded from participation to the study if she:

1. Has undergone breast radiation treatment and/or be preoperatively evaluated to require radiation treatment to the breast area during the course of the study.
2. Has collagen-vascular, connective tissue, or uncorrectable bleeding disorders as determined clinically by the PI.
3. Has a BMI that is ≥ 35.
4. Has any disease, including uncontrolled diabetes, which is clinically known to impact wound healing ability.
5. Has an autoimmune disease, an immune deficiency, or is on immune suppression drugs other than any other current treatment for breast cancer.
6. Currently has an alcohol/substance abuse problem or have had a relapse within 1 year prior to screening visit.
7. Is pregnant, or lactating.
8. Has concomitant unrelated condition of breast/chest wall/skin that, as determined by the PI, could affect the surgical outcome (e.g. significant chest wall abnormalities including pectus excavatum or pectus carinatum).
9. Has an abscess or infection at the time of surgery.
10. Has undergone previous breast surgery with the exception of breast biopsy, cyst removal, and lumpectomy.
11. Has had a prior soft tissue support device implanted in the breast or is participating in another clinical trial with a breast related device (e.g. drains, expanders, implants).
12. Has a known pork allergy or is sensitive to polysorbate.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Number of surgeries where a differentiation will be made between major and minor depending upon the requirement to enter the breast pocket under general anesthesia. | At month 36 post-implant placement
  Total numbers of major and of minor surgeries for each patient during the full trial period and including any surgeries that the PI determines are clinically still necessary at the end of the trial period. Major procedures are defined as those involving the patient to be treated in the OR: re-entering the implant pocket; soft-tissue flaps not performed under local anesthesia; general anesthesia; or procedures requiring inpatient admission. Other procedures, including for instance CT-guided percutaneous drainage or breast fat grafting (lipofilling), are defined as minor procedures.

SECONDARY OUTCOMES:
Post operative sensation at Postoperative | At Post-op Days 14, 30 and at Months 6, 12, 24, and 36 post implant placement
  Patients' subjective experience of sensation in the reconstructed breast as estimated by the subjective scale. In the experimental arm, this datum will be assessed at the POD 14 visit after the single stage implant (SSI) + ADM procedure; in the control arm\ this datum will be assessed at the POD 14 visit after the first stage and again POD 14 after the second surgical stage (TE/Implant exchange). The questionnaire will also be completed at Months 6, 12, 24 and 36.
Quality of life pre-operatively and at post operative | At month 6,12,24, and 36 post-implant placement
  Patients' QoL, including emotional and satisfaction status, will be assessed before the reconstruction procedure and at POD 30 after single stage implant (SSI) + ADM in the experimental group via the Short Form (SF)-36 questionnaire; and at POD 30 after TE/Implant exchange in the control group.

OTHER OUTCOMES:
Safety endpoints: evaluated by the number and type of complications that may occur. | At 6, 12, 24 and 36 months post-implant placement
  Safety will be assessed continuously for the study period.
Rate of capsular contracture at post operative | At month 6,12,24 and 36.
  The incidence of grade III and IV of Baker capsular contracture rates will be assessed after reconstruction.
Surgeon's evaluation of aesthetic outcome via photographs pre operatively | At month 6,12,24,and 36 post-implant placement
  Photographs, taken at follow up visits, will be assessed for aesthetic outcome after reconstruction. Conventional Anthropometric distance measurements will be assessed, including nipple-sternal notch, nipple-nipple and nipple-infra-mammary fold after reconstruction.
Costs related to in-hospital stay and devices. | At 6, 12, 24 and 36 months post-implant placement
  Overall cost of In-hospital stay (crude and including revision procedures) and device costs will be assessed.
Duration of post operative drainage. | At Post-op Day 30
  Duration of drain time from placement to removal and total drainage per day will be assessed after all surgical procedures where drains are used.
Total operating time | At Day of Surgery and Day of Expander/Implant exchange
  Operating time in minutes (in the control arm, operating time of the first and the second surgical stages will be recorded separately).
Acute inflammatory response | At Day of Discharge, Post-op Days 14 and 30
  Concatenated score as well as scores from each of the subscales will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Spano, MD, Principal Investigator — Fondazione IRCCS Instituto Nazionale dei Tumori
Locations (1):
- Fondazione IRCCS Instituto Nazionale dei Tumori, Milan, Italy